CLINICAL TRIAL: NCT03925480
Title: Preventing Young Infant Infections Using Azithromycin in Labour (PreYIAL): a Blinded, Randomised, Placebo-controlled Trial
Brief Title: Preventing Young Infant Infections Using Azithromycin in Labour (PreYIAL) Trial
Acronym: PreYIAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Ministry of Health, Fiji (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HREC 38057
Record Dates: First submitted 2019-04-04; First posted 2019-04-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Blinded, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matched drug and placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin (Experimental): A single 2g dose of Azithromycin
  Interventions: Drug: Azithromycin 500 mg Oral Tablet x 4
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Azithromycin 500 mg Oral Tablet x 4 — A single prophylactic dose of antibiotic given during labour
  Arms: Azithromycin
Drug: Matching Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
A trial to assess cumulative incidence of skin and soft tissue infections (SSTI) in infants (by three months of age) born to mothers receiving a single-dose of 2 grams of oral azithromycin during labour (or immediately prior to delivery in the case of caesarean section), compared to infants whose mothers received placebo.

DETAILED DESCRIPTION:
PreYIAL is a Phase III, double-blind, randomised, placebo controlled two arm trial of a single 2g dose of azithromycin or placebo, administered to women who have been admitted for delivery of their baby (either following onset of labour or for caesarean section).

The trial includes an estimated 2110 mothers/infant pairs (1055 per arm), with 12 months of follow-up for the mother/infant pair.

A swab-study within the main study involves 940 of the mother/infant pairs enrolled and involves follow-up for bacterial carriage outcomes, for 12 months.These swab-study participants will also be included in assessments of the infant and maternal microbiome.

ELIGIBILITY:
Inclusion criteria:

1. Pregnant women at least 18 years old intending to deliver at Colonial War Memorial Hospital (CWMH)
2. Women who have been admitted to CWMH for delivery at the time of eligibility assessment
3. Women who expect to be available, with their infant, for the duration of the study, and who agree to adhere to all protocol requirements
4. Women who will have a main place of residence within the Greater Suva area for the follow-up period and within a practical distance of the study site to allow compliance with protocol-required visits and follow-up, including attending follow-up at specified clinics
5. Women who have provided written informed consent prior to study-related procedures being performed

Exclusion criteria:

1. Women who have a known macrolide allergy
2. Women who have taken antibiotics in the week prior to randomisation
3. A women who is unable or unwilling to provide informed consent for her participation in the trial or the participation of her infant
4. Women who decide prior to randomisation that they are no longer willing to participate or to have their infant participate
5. Women who have ever received, or who are anticipated to receive during the study period, any investigational agent other than the study drug
6. Women who are CWMH, Murdoch Children's Research Institute (MCRI) or study site employees who work directly with study staff, or who are working on the study
7. Women taking warfarin due to the potential for drug interactions with azithromycin
8. Women with any cardiac abnormality
9. Women taking other medications known to prolong the QT interval such as antiarrhythmics; antipsychotic agents; antidepressants; and fluoroquinolones;
10. Women with known electrolyte disturbances: including in cases of hypokalaemia and hypomagnesaemia
11. Women who will undergo general anaesthetic for delivery
12. Women carrying a foetus with intrauterine death confirmed before randomisation
13. Women carrying a foetus with a prognosis unlikely to survive
14. Women with known HIV infection and/or taking nelfinavir
15. Women who have participated in the study during a previous pregnancy
16. Women who have been admitted for management of premature labour who have unruptured membranes (This is a temporary exclusion such that the participant may be assessed for eligibility again in the same or a subsequent admission to CWMH).
17. Women with renal impairment
18. Women with hepatic impairment
19. Women with myasthenia gravis
20. Women who are taking any ergot medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2110 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of skin and soft tissue infection by 3 months of age in infants | 3 months
  Born to mothers receiving a single dose of 2g Azithromycin during labour. Assessed by history and physical examination at 7 days, 6 weeks and 3 months.

SECONDARY OUTCOMES:
Cumulative incidence of skin and soft tissue infection, and other infections by 12 months of age in infants | Birth to 12 Months
  To compare intervention and placebo groups with regard to the cumulative incidence of infant infection (meningitis, sepsis, pneumonia, SSTI, fever, diarrhoea, urinary tract infection) up to 12 months of age;
Cumulative incidence of maternal infection by 6 weeks and 12 months post-delivery | Delivery to 12 months
  To compare intervention and placebo groups with regard to the cumulative incidence of maternal infection (mastitis, sepsis, post-operative wound infections, SSTI, fever, meningitis, pneumonia, abdominal or pelvic abscess, endometritis, urinary tract infection, pyelonephritis) by six weeks post-delivery, and similarly up to 12 months post-delivery
Cumulative incidence of antibiotic usage by 12 months in infants | Birth to 12 months
  To compare intervention and placebo groups with regard to the cumulative incidence of the number of courses of antibiotics prescribed to the infant up to 12 months of age;
Cumulative incidence of maternal antibiotic usage by 12 months post-delivery | Delivery to 12 months
  To compare intervention and placebo groups with regard to the cumulative incidence of the number of courses of antibiotics prescribed to the mother up to 12 months post-delivery
Number of infant participants with adverse events as assessed by adapted version of CTCAE v5.0 and DAID v2.1 | Birth to 12 months
  To compare the number of adverse events including solicited non serious adverse events and all serious adverse events as per study specific definitions throughout the duration of the study.
Number of maternal participants with adverse events as assessed by adapted version of CTCAE v5.0 and DAID v2.1 | Delivery to 12 months
  To compare the number of adverse events including solicited non serious adverse events and all serious adverse events as per study specific definitions throughout the duration of the study.
Number of infant and maternal participants with Staphylococcus aureus and/or Group A streptococcus as assessed by real-time quantitative PCR (qPCR) from impetigo swabs | Delivery/birth to 12 months
  The proportion of participants that have Staphylococcus aureus and/or Group A streptoccoccus detected by qPCR from impetigo swabs at key time points throughout the duration of the study, between the two groups
Number of infant and maternal participants with Staphylococcus aureus and/or Group A streptococcus with azithromycin nonsusceptibility cultured from impetigo swabs. | Delivery/birth to 12 months
  The proportion of participants that have Staphylococcus aureus and/or Group A streptococcus that is non susceptible to azithromycin cultured from impetigo swabs at key time points throughout the duration of the study, between the two groups
Swab study outcome - Prevalence of bacterial carriage as assessed by real-time quantitative PCR (qPCR) | Delivery/birth to 12 months
  Bacterial carriage, the proportion of participants that have at least one of the following bacterial species including GBS, SA, SPN, GAS or E. coli, assessed by qPCR at key time points throughout the duration of the study, between the two groups
Swab study outcome - Density of bacterial carriage as assessed by real-time quantitative PCR (qPCR) | Delivery/birth to 12 months
  Density of bacterial carriage, reported as log 10 genome equivalents/ml, of the participants that have at least one of the following bacterial species including GBS, SA, SPN, GAS or E. coli, assessed by qPCR at key time points throughout the duration of the study, between the two groups
Swab study outcome - Risk of maternal carriage identified through qPCR of common organisms relevant to Sexually Transmitted Infections (STI) | Delivery/birth to 6 months
  Maternal carriage of common organisms relevant to Sexually Transmitted Infections (STI) (including Chlamydia trachomatis, Neisseria gonorrhoeae, Trichomonas vaginalis, Mycoplasma genitalium, HSV-1 and HSV-2) as detected by qPCR at key time points throughout the duration of the study, between the two groups.
Swab study outcome - Risk of antibiotic nonsusceptibility in culture isolates | Delivery/birth to 12 months
  Antibiotic non susceptibility, based on the proportion of samples from mothers and infants that are non susceptible to antibiotics cultured in the two arms, at key time points throughout the duration of the study
Swab study outcome - The prevalence of infants with diagnoses that have been associated with microbiome dysbiosis | Delivery/birth to 6 months
  To compare the infant and maternal microbiome of specified body sites at key time points in the intervention and placebo groups

CONTACTS AND LOCATIONS:
Overall Officials: Fiona M Russell, BMBS PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Colonial War Memorial Hospital and Mother and Child Health Clinics, Suva, Central, Fiji

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the PreYIAL trial will be available six months after publication of the primary outcome.
  The study protocol, analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute by emailing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 6 months following publication of primary results for 15 years
Access Criteria: Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the DSMB must see and approve the analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgement and any additional costs involved must be covered. Data will only be shared with a recognised research institution which has approved the proposed analysis plan.

REFERENCES:
- [Background] Hume-Nixon M, Ratu T, Clark S, Nguyen CD, Neal EFG, Pell CL, Bright K, Watts E, Hart J, Mulholland K, Fong J, Rafai E, Sakumeni K, Tuibeqa I, Satzke C, Steer A, Russell FM. Prevention of young infant infections using oral azithromycin in labour in Fiji (Bulabula MaPei): study protocol of a randomised control trial. BMJ Open. 2022 Dec 1;12(12):e061157. doi: 10.1136/bmjopen-2022-061157. PMID 36456016
- [Result] Hume-Nixon M, Clark S, Ratu T, Nguyen CD, Neal EFG, Bright K, Strobel AG, Watts E, Hart J, Fong J, Rafai E, Sakumeni K, Steer A, Tuibeqa I, Russell FM. The safety and efficacy of a single dose of oral azithromycin given in labour to prevent skin and soft tissue infections in young infants in Fiji: a randomised controlled trial. BMC Med. 2025 Apr 28;23(1):246. doi: 10.1186/s12916-025-04070-6. PMID 40289086